CLINICAL TRIAL: NCT02636972
Title: The Progression From Dysmenorrhoea to Chronic Pelvic Pain: Investigation of the Role of Chronic Inflammatory Pain Phenotype in Peripheral Blood as a Potential Biomarker.
Brief Title: The Progression From Dysmenorrhoea to Chronic Pelvic Pain
Status: Completed | Type: Observational
Sponsor: University of Adelaide (Other)
Responsible Party: Principal Investigator, Dr Susan Evans, MBBS, FRANZCOG, FFPMANZCA, GAICD, University of Adelaide
Other Study IDs: PPAI-001
Record Dates: First submitted 2015-12-06; First posted 2015-12-22 (Estimated); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Dysmenorrhoea; Pelvic Pain; Chronic Pain
Keywords: TLR2; TLR4; Biomarker; TLR responsiveness; Peripheral blood responsiveness; Inflammatory pain
MeSH Terms: conditions — Dysmenorrhea; Pelvic Pain; Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood sample retained for future analysis (may include DNA analysis)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (7):
- Group 1: Mild or absent dysmenorrhoea and no other pelvic pain symptoms without contraceptive pill use.
- Group 2A: History of mild or absent dysmenorrhoea prior to pill use and no other pelvic pain symptoms with contraceptive pill use (Participants already using contraceptive pills).
  Interventions: Drug: OCPs
- Group 2B: History of severe dysmenorrhoea prior to pill use and no other pelvic pain symptoms with contraceptive pill use (Participants already using contraceptive pills).
  Interventions: Drug: OCPs
- Group 3: Severe dysmenorrhoea but without chronic pelvic pain and without contraceptive pill use.
- Group 4: Severe dysmenorrhoea but without chronic pelvic pain and with contraceptive pill use (Participants already using contraceptive pills).
  Interventions: Drug: OCPs
- Group 5: Chronic pelvic pain and severe dysmenorrhoea without contraceptive pill use
- Group 6: Chronic pelvic pain and severe dysmenorrhoea with contraceptive pill use (Participants already using contraceptive pills).
  Interventions: Drug: OCPs

INTERVENTIONS:
Drug: OCPs — Participants in the contraceptive pill groups can use any one of the following contraceptive pills:
  Oestradiol valerate and dienogest, drospirenone and ethinyl estradiol , ethinyloestradiol and levonorgestrel, cyproterone and ethinyl estradiol, ethinylestradiol and norethisterone, Nomegestrol Acetate and Oestradiol and Ethinyl Estra
  Groups: Group 2A; Group 2B; Group 4; Group 6

SUMMARY:
This is a cross-sectional observational study.

For participants resident in Adelaide, South Australia.

The study consists of 3 visits to the Pain and Anaesthesia Research Clinic (PARC), within the Royal Adelaide Hospital (RAH).

A total of 56 participants will be recruited for this study.

DETAILED DESCRIPTION:
The study will involve a screening visit followed by two visits to PARC for blood sampling and questionnaires.

At the baseline visit, blood samples to assess biomarkers and confirm hormonal status will be taken.

From screening until the final study visit a total of approximately 120 mL in blood samples will be taken from each participant.

The study aims to further knowledge in the presence of severe pelvic pain in young women which is an area that has been under-researched with regard to it's impact on society.

The study proposes to enroll 7 groups of 8 healthy nulliparous women aged 18-35 with the following characteristics:

Mild or absent dysmenorrhoea (pain scale 0-3) and no other pelvic pain symptoms. (3 groups)

* Group 1, without contraceptive pill use
* Group 2A , contraceptive pill user and with a history of mild or absent dysmenorrhoea prior to pill use
* Group 2B, contraceptive pill user and with a history of severe dysmenorrhoea (pain scale 7-10) prior to pill use

Severe dysmenorrhoea (pain scale 7-10), but without chronic pelvic pain. (2 groups)

* Group 3, without contraceptive pill use
* Group 4, contraceptive pill user

Chronic pelvic pain and severe dysmenorrhoea (2 groups)

* Group 5, without contraceptive pill use
* Group 6,contraceptive pill user

ELIGIBILITY:
Inclusion Criteria:

* Age between 16 to 35 years old

Exclusion Criteria:

* Irregular menstrual cycles
* Use of any reproductive hormonal preparations (other than the combined oral contraceptive pill), thyroxine, insulin or corticosteroids
* Presence of an inflammatory process, or clinically significant infection in the 4 weeks
* Clinically significant renal, hepatic, cardiac, auto-immune disease
* Current use of immunosuppressant medication such as hydroxychloroquine, methotrexate or azathioprine
* Inability to read or comprehend the written information provided
* Current use of medications known to affect TLR responsiveness including amitriptyline or minocycline
* Current use of any analgesics, including non-steroidal anti-inflammatory medications and opioids for 5 drug half-lives prior to the day of testing
* Current or previous pregnancy
* Body Mass index less than 18 or more than 30

Ages: 16 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Nulliparous women in good general health (can experience dysmenorrhoea (abscent, mild or severe), with or without pelvic pain and with or without contraceptive pill use)
Sampling Method: Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2014-11; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Reactivity of stimulated isolated peripheral blood immune cells | 2 weeks
  To determine if there are different inflammatory pain phenotypes between young women with either severe dysmenorrhoea alone, chronic pelvic pain from controls with mild or no dysmenorrhoea from the collected peripheral blood immune cells (assessed by cytokine output).

SECONDARY OUTCOMES:
Impact of pelvic pain on everyday activities using the Pelvic Pain Questionnaire | 2 weeks
  Secondary efficacy end point
Levels of anxiety and depression using the DAS21 | 2 weeks
  Secondary efficacy end point

CONTACTS AND LOCATIONS:
Overall Officials: Susan Evans, MBBS, Principal Investigator — PARC Research Clinic
Locations (1):
- PARC, Royal Adelaide Hospital, Adelaide, South Australia, Australia

IPD SHARING:
Plan to Share IPD: No